CLINICAL TRIAL: NCT05369650
Title: A Pilot Study on the Safety and Efficacy of Intravenous Infusion of Different Doses of Lidocaine for Postoperative Analgesia in Patients With Open Hepatectomy
Brief Title: To Explore the Safety and Efficacy of Intravenous Infusion of Different Doses of Lidocaine in Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Chunling Jiang, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-11
Record Dates: First submitted 2022-05-04; First posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Lidocaine; Injections

STUDY DESIGN:
Intervention Model Description: The experimental patients are randomly divided into three groups and received different doses of lidocaine and the control group received the same amount of saline.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants, the anesthesiologist, data collectors, the physicians performing the follow-up, and data analysts will be blinded to the group allocation. Blinding will maintain until the completion of the final analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lidocaine 1 group (Experimental): After induction of anesthesia, 1% lidocaine 1.5mg/kg (ideal body weight, 10min pumped) was injected intravenously with a micro pump, and then 1% lidocaine 1mg/kg.h (ideal body weight) was continuously pumped until the end of the operation , connected to patient-controlled intravenous analgesia (PCIA) pump containing lidocaine 0.3-1.5mg/kg.h after operation to 72h after operation.
  Interventions: Drug: Lidocaine Hydrochloride, Injectable
- Lidocaine 1.5 group (Experimental): After induction of anesthesia, 1% lidocaine 1.5mg/kg (ideal body weight, 10min pumped) was injected intravenously with a micro pump, and then 1% lidocaine 1.5mg/kg.h (ideal body weight) was continuously pumped until the end of the operation , connected to patient-controlled intravenous analgesia (PCIA) pump containing lidocaine 0.3-1.5mg/kg.h after operation to 72h after operation.
  Interventions: Drug: Lidocaine Hydrochloride, Injectable
- Lidocaine 2 group (Experimental): After induction of anesthesia, 1% lidocaine 1.5mg/kg (ideal body weight, 10min pumped) was injected intravenously with a micro pump, and then 1% lidocaine 2mg/kg.h (ideal body weight) was continuously pumped until the end of the operation , connected to patient-controlled intravenous analgesia (PCIA) pump containing lidocaine 0.3-1.5mg/kg.h after operation to 72h after operation.
  Interventions: Drug: Lidocaine Hydrochloride, Injectable

INTERVENTIONS:
Drug: Lidocaine Hydrochloride, Injectable — The lidocaine group 1, 1.5 and 2 groups were injected with 1% lidocaine 1.5mg/kg (ideal body weight, 10min infusion) after anesthesia induction, respectively, and then continued to infuse 1% lidocaine. 1mg/kg.h, 1.5mg/kg.h, 2mg/kg.h (ideal body weight) until the end of the operation, and a patient-controlled intravenous analgesia (PCIA) pump containing lidocaine (PCIA) 0.3-1.5mg/kg after surgery. h to 72h after surgery.

SUMMARY:
All patients who met the inclusion criteria were randomly divided into four groups, 30 cases in each group, which were lidocaine group 1, lidocaine group 1.5, lidocaine group 2, and the placebo group In lidocaine group 1, lidocaine group 1.5, and lidocaine group 2, 1% lidocaine 1.5 mg/kg was intravenously infused with a micropump after anesthesia induction, and the infusion was completed within 10 minutes according to the ideal body weight, and then continued for 1% lidocaine was infused at 1 mg/kg.h, 1.5 mg/kg.h and 2 mg/kg.h respectively until the end of the operation. In the placebo group, the same volume of normal saline was used instead.

DETAILED DESCRIPTION:
All patients who met the inclusion criteria were randomly divided into four groups, 30 cases in each group, which were lidocaine group 1, lidocaine group 1.5, lidocaine group 2, and the placebo group In lidocaine group 1, lidocaine group 1.5, and lidocaine group 2, 1% lidocaine 1.5 mg/kg was intravenously infused with a micropump after anesthesia induction, and the infusion was completed within 10 minutes according to the ideal body weight, and then continued for 1% lidocaine was infused at 1 mg/kg.h, 1.5 mg/kg.h and 2 mg/kg.h respectively until the end of the operation. In the placebo group, the same volume of normal saline was used instead.Postoperative pain management during the first 72 postoperative hours will involve the use of a PCIA device, which will contain lidocaine 30mg/kg, sufentanil 2 μg/kg, granisetron 12 mg diluted to 200 mL in 0.9 % normal saline. In the placebo group, the same volume of normal saline will be administered during anesthesia. The postoperative PCIA device will contain sufentanil 2 μg/kg, granisetron 12 mg diluted to 200 mL in 0.9% normal saline solution with a total volume of 200 ml. All the background infusions of PCIA will set at 2 ml/h, the bolus volume of each PCIA press is 2 ml and the lockout interval is 15 min.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70 years old
* American Society of Anesthesiologists(ASA) Ⅰ～III
* BMI≤30
* Intended for open liver resection Exclusion criteria：1. Long-term opioid users 2. Patients with contraindications or allergies to any drugs (lidocaine, etc.) used in this study 3. Patients with severe hepatic insufficiency before surgery (defined as total bilirubin>1.46mg/dl), renal insufficiency (glomerular filtration rate <30ml/min/1.73m2 or end-stage renal disease) 4. Associated with severe heart disease (second or third degree atrioventricular block); severe heart failure (ejection fraction <50%); sinus bradycardia; patient 6. Patients who participated in other clinical trials within 3 months before enrollment in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-07-27 (Actual); Primary Completion 2022-05-27 (Estimated); Study Completion 2022-09-27 (Estimated)

PRIMARY OUTCOMES:
Immediate postoperative plasma lidocaine concentration | Immediately after surgery
  Plasma lidocaine concentration is an important indicator for evaluating the safety of the drug during use

SECONDARY OUTCOMES:
Plasma lidocaine concentration immediately after loading | 30 minutes before surgery
  Plasma lidocaine concentration is an important indicator for evaluating the safety of the drug during use
24-hour postoperative plasma lidocaine concentration | 24-hour postoperative
  Plasma lidocaine concentration is an important indicator for evaluating the safety of the drug during use
The incidence of lidocaine toxicity within 72 hours after operation | within 72 hours after operation
  Lidocaine toxicity mainly includes neurological manifestations such as dizziness, tinnitus, convulsions, cardiac manifestations such as bradycardia, new severe atrioventricular block and so on.
The incidence of moderate to severe pain at 24、48 and 72 hours after surgery at rest and during movement; | 24，48 and 72 hours after surgery
  he pain is evaluated using numerical rating scale（NRS). NRS scores range from 0 to 10 points, with 0 points representing no pain, 1-3 points representing mild pain, 4-6 points representing moderate pain, 7-9 points representing severe pain and 10 points representing the strongest pain.
The cumulative morphine consumption at 24, 48 and 72 hours postoperatively | At the end of the surgery，24，48 and 72 hours after surgery
  intra-operative and postoperative opioid use is reported as morphine milligram
Bowel function recovery | At 3 days after surgery
  defined as the time to first defecation or time to first flatus
Postoperative hospital stay | up to 30 days
  The days of hospital stay after the operation were calculated from the first day after the operation to the days of discharge.
Patient satisfaction scores | 72 hours after surgery
  (satisfaction scores regarding pain control and the overall recovery process were obtained at 72 hours after surgery, using a 11-point Likert scale, with 0 indicating "very dissatisfied"and10 indicating "very satisfied"

CONTACTS AND LOCATIONS:
Overall Officials: Chunling Jiang, PhD, Study Director — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No